CLINICAL TRIAL: NCT07390474
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of the V2 Apex-Directed Immunogens DV201P-RNA and DV202B1-RNA in Adult Participants Without HIV
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of the V2 Apex-Directed Immunogens DV201P-RNA and DV202B1-RNA in Adult Participants Without HIV
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 322
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HIV
Keywords: Healthy Participants; HIV Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: 50 mcg (Experimental): DV201P-RNA (50 mcg) at weeks 0 and 12.
  Followed by:
  DV202B1-RNA (50 mcg) at weeks 24 and 40.
  Interventions: Biological: DV201P-RNA; Biological: DV202B1-RNA
- Group 2: 100 mcg (Experimental): DV201P-RNA (100 mcg) at weeks 0 and 12.
  Followed by:
  DV202B1-RNA (100 mcg) at weeks 24 and 40.
  Interventions: Biological: DV201P-RNA; Biological: DV202B1-RNA
- Group 3: 150 mcg (Experimental): DV201P-RNA (150 mcg) at weeks 0 and 12.
  Followed by:
  DV202B1-RNA (150 mcg) at weeks 24 and 40.
  Interventions: Biological: DV201P-RNA; Biological: DV202B1-RNA
- Group 4: TBD* (Experimental): DV202B1-RNA (50 mcg or 100 mcg or 150 mcg; highest dose that is determined to be safe and well tolerated from Groups 1-3) at weeks 0 and 12.
  Interventions: Biological: DV202B1-RNA

INTERVENTIONS:
Biological: DV201P-RNA — To be administered intramuscularly as a split dose.
  Arms: Group 1: 50 mcg; Group 2: 100 mcg; Group 3: 150 mcg
Biological: DV202B1-RNA — To be administered intramuscularly as a split dose.

SUMMARY:
This is a phase 1, multicenter, open-label, dose escalation, first-in-human (FIH) trial to evaluate the safety and immunogenicity of DV201P-RNA and DV202B1-RNA, immunogens designed to induce HIV-1 envelope (Env) V2 apex-specific broadly neutralizing antibodies (V2 apex bnAbs). Both vaccines consist of a modified mRNA encapsulated in lipid nanoparticles (LNP) that when translated in cells produces HIV-1 Env gp150 transmembrane trimers. The trial will enroll adult volunteers without HIV and in overall good health.

ELIGIBILITY:
Inclusion Criteria:

1. Demonstrates an understanding of the study and is able and willing to complete the informed consent process.
2. At least 18 years old at screening and up to 55 years old on day of enrollment.
3. Available for clinic follow-up through the last clinic visit.
4. Willing to undergo study procedures as outlined in the schedule of procedures (Appendix A).
5. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 322 PSRT are required prior to enrollment into HVTN 322.
6. In good general health according to the clinical judgment of the site investigator.
7. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgment of the site investigator.
8. Agrees to discuss their potential for HIV acquisition and agrees to HIV prevention counseling.
9. Hemoglobin (Hgb):

   * 11.0 g/dL for women
   * 13.0 g/dL for men
10. White blood cell (WBC) count of 2,500 to 12,000/mm3. WBC over 12,000/mm3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted.
11. Platelet count of 125,000 to 550,000/mm3.
12. Alanine aminotransferase (ALT) <2.5× the upper limit of institutional reference range.
13. Serum creatinine ≤1.1× the upper limit of normal (ULN) based on the institutional normal range.
14. Total measured serum calcium level >8.5 mg/dL.
15. Systolic blood pressure of 90 to <140 mm Hg and diastolic blood pressure of 50 to <90 mm Hg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mm Hg systolic and 90 mmHg diastolic. A single measurement of ≥160 mm Hg systolic or ≥100 mm Hg diastolic during the current study evaluation is exclusionary.
16. HIV test results by one of the following options:

    • Negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA) or

    • Negative results on two different brands of HIV rapid tests (one of which must be FDA-approved)
17. Negative for anti-Hepatitis C virus (HCV) Abs or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
18. Negative for Hepatitis B surface antigen (Ag).
19. For women of pregnancy potential:

    • Must agree to use effective means of contraception from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint (see Appendix D).

    • Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.

    Note: Women who have had a total hysterectomy, bilateral oophorectomy, or bilateral salpingectomy (verified by medical records) or menopause (no menses for ≥1 year) are not required to undergo pregnancy testing.
20. Women of pregnancy potential must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Women who are breastfeeding or pregnant.
2. Body mass index (BMI) ≥40. Enrollment of individuals with BMI ≥40 who are in good health, as assessed by the site investigator, may be considered by PSRT approval.
3. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤8% within the last 6 months (sites may draw these at screening).
4. Previous or current recipient of an investigational HIV vaccine (previous placebo/control recipients are not excluded).
5. Receipt of non-HIV investigational vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
6. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use or prednisone dose of ≥10 mg/day, within 3 months prior to enrollment.
7. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
8. Receipt of any of the following within 4 weeks prior to enrollment:

   • Live replicating vaccine

   • Any mRNA-based vaccine with FDA licensure, FDA EUA, or WHO EUL

   • ACAM2000 vaccine >28 days prior with a vaccination scab still present
9. Receipt of any vaccine that is not covered in exclusion criterion #8 within 14 days prior to enrollment. Please note this includes replication-incompetent vaccines such as the Jynneos vaccine for the prevention of mpox (formerly known as monkeypox) disease.
10. History of myocarditis and/or pericarditis.
11. Initiation of Ag-based immunotherapy for allergies within the past year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
12. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. (Receipt of an investigational research agent with a half-life of 7 or fewer days more than 4 weeks prior to enrollment is not exclusionary.) If a potential participant has received investigational agents with a half-life of more than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
13. History of serious reaction (eg, hypersensitivity, anaphylaxis) to any mRNA vaccine, including Comirnaty (Pfizer) and Spikevax (Moderna), or to any drug administered systemically as a polyethylene glycol containing LNP, including doxorubicin (Doxil, Caelyx, ThermoDox), cisplatin (Lipoplatin), and irinotecan (Onivyde).
14. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
15. Urticarial episode (idiopathic or known etiology) within the past year.
16. History of chronic urticaria.
17. History of urticaria previously associated with immunization.
18. Bleeding disorder diagnosed by a clinician that would make study procedures a contraindication.
19. History of seizure(s) within the past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
20. Asplenia or functional asplenia.
21. Active duty and reserve US military personnel.
22. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, including but not limited to clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, any suicide attempt within the past year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgment of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
23. Asthma is excluded if the participant meets any of the following criteria:

    • Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year

    • Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would not exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma)

    • Uses a short-acting rescue inhaler more than 2 days per week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity)

    • Uses medium- to high-dose inhaled corticosteroids (>250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA])

    • Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
24. A participant with a history of a PIMMC, either active or remote. Specific examples are listed in Appendix E (AESI index). Not exclusionary: (1) remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms; (2) mild psoriasis or other mild, uncomplicated, localized, or dermatologic condition that does not require ongoing systemic treatment; (3) remote history (>10 years ago) of Kawasaki disease without sequelae; (4) celiac disease well controlled for 6 months with diet only.
25. History of allergy to local anesthetic (Novocaine, Lidocaine).
26. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-12-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Local reactogenicity for a minimum of 14 days following receipt of any study vaccine | Day 0 (vaccination) through 14 days post-vaccination; at days 15, 99, 183, and 295
Systemic reactogenicity for a minimum of 14 days following receipt of any study vaccine | Day 0 (vaccination) through 14 days post-vaccination; at days 15, 99, 183, and 295
Serious adverse events (SAEs), medically attended AEs (MAAEs), AEs of special interest (AESIs), and AEs leading to withdrawal/discontinuation collected throughout study; additionally, all AEs collected for 30 days after receipt of any study vaccination | From informed consent through end of study for SAEs, MAAEs, AESIs, and AEs leading to withdrawal/discontinuation; all AEs for 30 days after receipt of any study vaccination
Response rate of V2 apex-specific IgG+ B cells as assessed by flow cytometry 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Frequency of V2 apex-specific IgG+ B cells as assessed by flow cytometry 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Response rate of differential serum Ab neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses, as measured by the TZM-bl assay at 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Magnitude of differential serum Ab neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses, as measured by the TZM-bl assay at 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Response rate of serum IgG binding antibodies to autologous HIV Env stabilized trimers, as assessed by binding antibody multiplex assay (BAMA) at 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Magnitude of serum IgG binding antibodies to autologous HIV Env stabilized trimers, as assessed by BAMA at 2 weeks after second vaccination | 2 weeks after the second vaccination (Day 99)
Response rate of differential serum Ab neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses as measured by TZM-bl pseudovirus assay 2 weeks after the third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)
Magnitude of differential serum Ab neutralization of precursor detection viruses and corresponding epitope knock-out mutant forms of the viruses as measured by TZM-bl pseudovirus assay 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)

SECONDARY OUTCOMES:
Response rate of serum IgG binding to HIV Env-stabilized trimers as assessed by BAMA at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)
Magnitude of serum IgG binding to HIV Env-stabilized trimers as assessed by BAMA at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)
V2 specificity of serum IgG binding to HIV Env-stabilized trimers as assessed by BAMA at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)
Breadth of serum IgG binding to HIV Env-stabilized trimers as assessed by BAMA at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination (Days 183 and 295)
Response rate of V2 apex-specific IgG+ B cells as assessed by flow cytometry at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination
Frequency of V2 apex-specific IgG+ B cells as assessed by flow cytometry at 2 weeks after third and fourth vaccinations (Groups 1-3) | 2 weeks after the third vaccination and 2 weeks after the fourth vaccination
Frequency of V2 apex broadly neutralizing antibody (bnAb) lineage sequences as measured by B-cell receptor (BCR) single cell sequencing of V2 apex-specific IgG+ B cells | 2 weeks after the fourth vaccination for Groups 1-3; 2 weeks after the second vaccination for Group 4
Epitope-specific response rates as measured by EMPEM at 2 weeks after vaccination | 2 weeks after the fourth vaccination for Groups 1-3; 2 weeks after the second vaccination for Group 4
Response rate of serum antibody neutralization of heterologous HIV-1 strains as measured by TZM-bl assay at 2 weeks after vaccination | Groups 1-3: 2 weeks after the second vaccination and 2 weeks after the fourth vaccination, Group 4: 2 weeks after the second vaccination
Magnitude of serum antibody neutralization of heterologous HIV-1 strains as measured by TZM-bl assay at 2 weeks after vaccination | Groups 1-3: 2 weeks after the second vaccination and 2 weeks after the fourth vaccination, Group 4: 2 weeks after the second vaccination

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - The Ponce de Leon Center CRS, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Research Center; Emory University, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No